CLINICAL TRIAL: NCT02329600
Title: Evaluation of Systemic Administration of Green Tea Polyphenols as a Supportive Antioxidant Agent in the Management of Oral Lichen Planus
Brief Title: Evaluation of Green Tea as Antioxidant Agent in Management of Oral Lichen Planus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of periodontology and Oral Medicine, faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: polyphenol_TOC_OLP
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-09

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Tea; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control subjects (No Intervention): 10 systemically healthy control subjects taking no medication.
- OLP and corticosteroid (Active Comparator): 15 Patients who were previously diagnosed with oral lichen planus presented in acute exacerbation were treated with topical corticosteroids; Triamcinolone acetonide (Kenalog in orabase: Bristol-Myers, Squibb, Spain) applied topically 4 times a day i.e. following each meal and at bed time for one month.
  Interventions: Drug: Triamcinolone Acetonide
- OLP and corticosteroid and green tea (Experimental): 15 Patients who were previously diagnosed with oral lichen planus presented in acute exacerbation were treated with both topical corticosteroids; Triamcinolone acetonide (Kenalog in orabase: Bristol-Myers, Squibb, Spain) applied topically 4 times a day i.e. following each meal and at bed time for one month in addition to green tea tablets 200 mg (Green tea extract 5:1, El Obour For Modern Pharmaceutical Industries) as one tablet a day also for one month.
  Interventions: Drug: green tea tablets (Green tea extract 5:1) 200 mg; Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: green tea tablets (Green tea extract 5:1) 200 mg — Green tea is a product made from the Camellia sinensis plant. The fresh leaves are used to make medicine. the green tea extract is presented in a form of tablets 200 mg and is taken orally.
  Other Names: Green Tea Polyphenolic Fraction
  Arms: OLP and corticosteroid and green tea
Drug: Triamcinolone Acetonide — topical corticosteroids (Kenalog in orabase: Bristol-Myers, Squibb, Spain) applied topically 4 times a day i.e. following each meal and at bed time for one month
  Other Names: Kenalog in orabase
  Arms: OLP and corticosteroid; OLP and corticosteroid and green tea

SUMMARY:
The study included forty individuals divided into 3 groups. 10 control subjects, 15 oral lichen planus (OLP) patients who were treated with topical corticosteroids and 15 oral lichen planus (OLP) patients who were treated with topical corticosteroids and green tea tablets.

DETAILED DESCRIPTION:
This study included forty individuals divided into 3 groups. Group A; 10 systemically healthy control subjects not receiving medication.

Group B; 15 Patients who were previously diagnosed with OLP presented in acute exacerbation were treated with topical corticosteroids; Triamcinolone acetonide (Kenalog in orabase: Bristol-Myers, Squibb, Spain) applied topically 4 times a day i.e. following each meal and at bed time for one month.

Group C; 15 Patients who were previously diagnosed with OLP presented in acute exacerbation were treated with both topical corticosteroids; Triamcinolone acetonide (Kenalog in orabase: Bristol-Myers, Squibb, Spain) applied topically 4 times a day i.e. following each meal and at bed time for one month in addition to green tea tablets 200 mg (Green tea extract 5:1, El Obour For Modern Pharmaceutical Industries) as one tablet a day also for one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with painful oral lichen planus lesions
* Free of any visible oral lesions other than oral lichen planus
* Free of any systemic diseases

Exclusion Criteria:

* Topical treatment or systemic therapy of OLP for one month before starting the study
* Pregnant or breast feeding women
* Smokers
* Use of corticosteroids or other immunosuppressive drugs

Ages: 30 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noha Ghallab, M.D., Study Chair — Associate Professor of periodontology and Oral Medicine faulty of oral and dental medicine Cairo Unv.; Enji Ahmed, M.D., Study Director — Lecturer of periodontology and Oral Medicine faulty of oral and dental medicine Cairo Unv.; Ghada Nabil, B.D.S, Principal Investigator — Instructor of periodontology and Oral Medicine faulty of oral and dental medicine Cairo Unv.

REFERENCES:
- [Result] Agha-Hosseini F, Mirzaii-Dizgah I, Farmanbar N, Abdollahi M. Oxidative stress status and DNA damage in saliva of human subjects with oral lichen planus and oral squamous cell carcinoma. J Oral Pathol Med. 2012 Nov;41(10):736-40. doi: 10.1111/j.1600-0714.2012.01172.x. Epub 2012 May 15. PMID 22582895
- [Result] Nakagawa T, Yokozawa T. Direct scavenging of nitric oxide and superoxide by green tea. Food Chem Toxicol. 2002 Dec;40(12):1745-50. doi: 10.1016/s0278-6915(02)00169-2. PMID 12419687
- [Result] Sander CS, Cooper SM, Ali I, Dean D, Thiele JJ, Wojnarowska F. Decreased antioxidant enzyme expression and increased oxidative damage in erosive lichen planus of the vulva. BJOG. 2005 Nov;112(11):1572-5. doi: 10.1111/j.1471-0528.2005.00743.x. PMID 16225582
- [Result] Singh BN, Shankar S, Srivastava RK. Green tea catechin, epigallocatechin-3-gallate (EGCG): mechanisms, perspectives and clinical applications. Biochem Pharmacol. 2011 Dec 15;82(12):1807-21. doi: 10.1016/j.bcp.2011.07.093. Epub 2011 Jul 30. PMID 21827739
- [Result] Zhang J, Zhou G. Green tea consumption: an alternative approach to managing oral lichen planus. Inflamm Res. 2012 Jun;61(6):535-9. doi: 10.1007/s00011-012-0440-z. Epub 2012 Feb 10. PMID 22322481

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Subjects | OLP and Corticosteroid | OLP and Corticosteroid and Green Tea
Started | 10 | 15 | 15
Completed | 10 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Subjects | OLP and Corticosteroid | OLP and Corticosteroid and Green Tea | Total
Number analyzed (Participants) | 10 | 15 | 15 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 15 | 40
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (2.7) | 41.4 (9.7) | 44.3 (16.2) | 38 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 9 | 24
  Male | 5 | 5 | 6 | 16
Region of Enrollment [Number; unit: participants]
  Egypt | 10 | 15 | 15 | 40

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: pain was assessed by visual analogue scale (1-10) 1 indicates better and 10 worse, 1 month after treatment
Time Frame: one month after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Subjects | OLP and Corticosteroid | OLP and Corticosteroid and Green Tea
Number analyzed (Participants) | 10 | 15 | 15
units on a scale | 0 (0) | 4 (2.4) | 4.4 (2.1)

2. Secondary Outcome: Salivary Total Oxidative Capacity
Description: total oxidative capacity was assessed in whole unstimulated saliva by ezyme-linked immunosorbent assay (umol/L) at 1 month after treatment
Time Frame: one month after treatment
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Control Subjects | OLP and Corticosteroid | OLP and Corticosteroid and Green Tea
Number analyzed (Participants) | 10 | 15 | 15
umol/L | 6.37 (4.06) | 58.41 (16.3) | 23.27 (12.95)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Subjects | OLP and Corticosteroid | OLP and Corticosteroid and Green Tea
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/10 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No